CLINICAL TRIAL: NCT04854590
Title: IMFINZI® Injection 120 mg, 500 mg Specific-Clinical Experience Investigation in Patients With Extensive Stage Small Cell Lung Cancer
Brief Title: IMFINZI Study in Patients With Extensive Stage Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D419QC00006
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Carcinoma, Small Cell
MeSH Terms: conditions — Carcinoma, Small Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Weeks

SUMMARY:
To capture safety(FN) when IMF is administered to patients with extensive stage small cell lung cancer in clinical practice after launch

DETAILED DESCRIPTION:
To capture the onset (incidence, severity, intervention, outcome, and others) of febrile neutropenia in patients with extensive stage small cell lung cancer who receive durvalumab in combination with platinum agent and etoposide under the actual use.

ELIGIBILITY:
Inclusion Criteria:

-Patients with extensive stage small cell lung cancer who are receiving the product in combination with platinum agent and etoposide.

Exclusion Criteria:

-Patients who have no treatment history with the product (i.e.,durvalumab)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with extensive stage small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Incidence of febrile neutropenia (yes/no) and by severity (CTCAE grade) | 16weeks

CONTACTS AND LOCATIONS:
Overall Officials: Toshimitsu Tokimoto, Study Director — Astrazeneca KK
Locations (18):
- Japan (18):
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Gunma
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Kanagawa
  - Research Site, Miyagi
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Saitama
  - Research Site, Shizuoka
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Wakayama

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419QC00006&attachmentIdentifier=91647536-400f-44bc-9088-a2bac5b09a8f&fileName=Synopsis_for_D419QC00006.pdf&versionIdentifier=